CLINICAL TRIAL: NCT02070146
Title: Prospective Data Collection Initiative on Colorectal Cancer - a Prospective Observational Cohort Study -
Brief Title: Prospective Data Collection Initiative on Colorectal Cancer
Acronym: PLCRC
Status: Recruiting | Type: Observational
Sponsor: Dutch Colorectal Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: 12-510
Record Dates: First submitted 2013-08-07; First posted 2014-02-25 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Blood and tumor tissue will be stored.
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Survival after colorectal cancer (CRC) diagnosis strongly depends on local tumor extent, lymph node involvement and the presence of distant metastases. However, there remains great inter-patient variability regarding treatment outcome. A combination of biochemical factors, histopathological features, genomic profile, environmental factors and other clinical factors are likely to influence prognosis and treatment effect, independent from tumor stage, but it is still unclear which, how, and to what extent these factors can influence tumor recurrence and mortality in both early stage (I-III) and late stage (IV) CRC, small bowel cancer and anal cancer.

Although the results from prospective clinical trials will remain the backbone of evidence based medicine, this concerns a highly selected patient population since the large majority (85%-95%) of cancer patients do not participate in clinical trials for various reasons. It is unlikely that trial participation will significantly improve in the near future. This fact has the following implications: 1) It is highly desirable to validate the results from trials in the general patient population. However, this is complicated by the fact that the documentation of patients treated in general practice (i.e. outside the scope of clinical trials) is largely insufficient to provide comparable patient cohorts in terms of prognostic characteristics and treatment parameters. 2) There is an increased availability of novel technologies that provide molecular markers with potential prognostic and/or predictive value. To test the clinical value of these markers large numbers of patients are required which greatly exceeds the number of patients who consent to participate in prospective clinical trials. 3) as a result of rapid technical developments, a range of new minimally invasive treatment options are entering the market. These interventions have the potential to be of great benefit for patients in terms of improved local control, higher probability of complete tumor removal, less damage to surrounding tissue, faster recovery and less short and long term side effects. Still, the interventions will have to prove their effectiveness, safety and superiority (or non-inferiority) to standard cancer treatments on a patient level. A prospective observational cohort study has the great opportunity to fill this gap.

DETAILED DESCRIPTION:
Objectives

* To start a prospective observational cohort study of CRC, small bowel and anal cancer patients from their primary diagnosis until death.
* After obtaining Informed Consent, to prospectively collect data on medical history, comorbidities, baseline clinical parameters, imaging results, pathology results, tumor characteristics, treatment, treatment outcomes, hospital stays, interventions and (S)AEs.
* After obtaining separate Informed Consent for collecting data on health related quality of life and work ability, to collect data on patient reported outcome measures.
* After obtaining separate Informed Consent, to collect blood, (tumor) tissue or other body material, obtained during routine practice, for observational studies or storage in the biobank.
* The cohort will serve as an infrastructure geared towards efficient, safe and comprehensive clinical evaluation of new interventions for patients with CRC according to the Trials within Cohorts (TwiCs) design.

Expected outcome

* More accurate data on the treatment and clinical and patient reported outcomes of CRC, small bowel and anal cancer in daily practice.
* A continuous infrastructure for a large variety of research purposes including:

A. Prognostic and predictive research. B. Molecular research and (epi)genetic research. C. Comparison of new interventions for patients with CRC, small bowel and anal cancer according to the Trials within Cohorts (TwiCs) design. D. Health care policies and cost-effectiveness studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological proof of colorectal, small bowel and anal cancer, or a strong suspicion after imaging.
* Informed consent for longitudinal observational data collection.

Exclusion Criteria:

* Mentally incompetent patients.

Participation of patients to the PLCRC project does not exclude participation in any other ongoing or future study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with colorectal, small bowel and anal cancer, who are recently diagnosed, have a strong suspicion without pathological confirmation or are currently under treatment or follow up in one of the participating hospitals will be asked to participate in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2051-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 10 years

SECONDARY OUTCOMES:
Health related quality of life | 3, 6, 12, 24, 36, 48 months
  measured by EORTC QLQ questionnaire
Grade 3/4 (serious) adverse events | 3 months
Disease free survival | up to 10 years
Overall survival | up to 10 years
Work Ability Index (WAI) | 3, 6, 12, 24, 36, 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Koopman, MD, PhD, Principal Investigator — UMC Utrecht
Locations (67):
- Netherlands (67):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - Antoni van Leeuwenhoek, Amsterdam
  - OLVG, Amsterdam
  - VUmc, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Wilhelmina Ziekenhuis Assen, Assen
  - Maasziekenhuis Pantein, Beugen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia ziekenhuis, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf, Delft
  - Deventer Ziekenhuizen, Deventer
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Anna Ziekenhuis, Geldrop
  - Admiraal De Ruyter Ziekenhuis, Goes
  - Rivas Beaterix Ziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - UMC Groningen, Groningen
  - Spaarne Gasthuis, Haarlem
  - Saxenburgh Groep, Hardenberg
  - St.Jansdal, Harderwijk
  - Frisius MC Heerenveen, Heerenveen
  - Elkerliek Ziekenhuis, Helmond
  - Ziekenhuisgroep Twente, Hengelo
  - Tergooi, Hilversum
  - Treant Zorggroep, Hoogeveen
  - Dijklander Ziekenhuis, Hoorn
  - Frisius MC Leeuwarden, Leeuwarden
  - Alrijne, Leiden
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht UMC+, Maastricht
  - MAASTRO, Maastricht
  - St. Antonius ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud UMC, Nijmegen
  - Bernhoven, Oss
  - Laurentius Ziekenhuis, Roermond
  - Bravis ziekenhuis, Roosendaal
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Zuyderland Medisch Centrum, Sittard
  - Antonius Ziekenhuis, Sneek
  - ZorgSaam, Terneuzen
  - Haaglanden MC, The Hague
  - HagaZiekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - St. Jans Gasthuis, Weert
  - Zaans Medisch Centrum, Zaandam
  - Isala, Zwolle

REFERENCES:
- [Derived] Smit KC, Derksen JWG, Stellato RK, VAN Lanen AS, Wesselink E, Belt EJT, Balen MC, Coene PPLO, Dekker JWT, DE Groot JW, Haringhuizen AW, VAN Halteren HK, VAN Heek TT, Helgason HH, Hendriks MP, DE Hingh IHJT, Hoekstra R, Houtsma D, Janssen JJB, Kok N, Konsten JLM, Los M, Meijerink MR, Mekenkamp LJM, Peeters KCMJ, Polee MB, Rietbroek RC, Schiphorst AHW, Schrauwen RWM, Schreinemakers J, Sie MPS, Simkens L, Sonneveld EJA, Terheggen F, Iersel LV, Vles WJ, Wasowicz-Kemps DK, DE Wilt JHW, Kok DE, Winkels RM, Kampman E, VAN Duijnhoven FJB, Koopman M, May AM. Determinants of Physical Activity among Patients with Colorectal Cancer: From Diagnosis to 5 Years after Diagnosis. Med Sci Sports Exerc. 2024 Apr 1;56(4):623-634. doi: 10.1249/MSS.0000000000003351. Epub 2023 Nov 27. PMID 38079324